CLINICAL TRIAL: NCT02647359
Title: A Phase 2, Multicenter, Randomized, Double-Masked, Placebo-Controlled Study of the Safety and Efficacy of Ataluren (PTC124) for the Treatment of Nonsense Mutation Aniridia
Brief Title: Study of Ataluren in Participants With Nonsense Mutation Aniridia
Acronym: STAR
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: PTC Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PTC124-GD-028 ANI
Record Dates: First submitted 2015-12-29; First posted 2016-01-06 (Estimated); Results first posted 2022-05-27 (Actual); Last update posted 2022-05-27 (Actual); Status verified 2022-04

CONDITIONS: Aniridia
MeSH Terms: conditions — Aniridia | interventions — ataluren

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Ataluren (Experimental): Participants will receive ataluren orally 3 times a day (TID) at a dose of 10 milligrams per kilogram (mg/kg) in the morning, 10 mg/kg at midday, and 20 mg/kg in the evening for 48 weeks in Stage 1 (double-masked period) and for additional 96 weeks in Stage 2 (open-label extension period). Participants, who complete Stage 2 and agree to continue in open-label sub-study, will continue to receive ataluren treatment at same dose as mentioned above, for 96 weeks or until commercial availability of ataluren for this indication, whichever is first, or until a positive risk-benefit assessment in this indication is not demonstrated.
  Interventions: Drug: Ataluren
- Placebo (Placebo Comparator): Participants will receive placebo matching to ataluren TID orally in the morning, at midday, and in the evening for 48 weeks in Stage 1 (double-masked period) and ataluren orally TID at a dose of 10 mg/kg in the morning, 10 mg/kg at midday, and 20 mg/kg in the evening for additional 96 weeks in Stage 2 (open-label extension period). Participants, who complete Stage 2 and agree to continue in open-label sub-study, will continue to receive ataluren treatment at same dose as mentioned above, for 96 weeks or until commercial availability of ataluren for this indication, whichever is first, or until a positive risk-benefit assessment in this indication is not demonstrated.
  Interventions: Drug: Ataluren; Drug: Placebo

INTERVENTIONS:
Drug: Ataluren — Ataluren oral suspension will be administered as per the dose and schedule specified in the respective arms.
  Other Names: PTC124; Translarna
Drug: Placebo — Placebo will be administered as per the schedule specified in the respective arm.
  Arms: Placebo

SUMMARY:
This study is designed to evaluate the effect of ataluren on Maximum Reading Speed as measured using the Minnesota Low Vision Reading Test (MNREAD) Acuity Charts in participants with nonsense mutation aniridia. This study involves a 4-week screening period, a 144-week treatment period (Stage 1: Weeks 1 to 48 [double-masked treatment] and Stage 2: Weeks 49 to 144 [open label treatment]), an optional 96-week open label extension sub-study, and a 4-week post-treatment follow-up period (either study completion or early termination). Participants that choose not to participate in the sub-study will be required to complete the post-treatment follow-up visit at the end of the Stage 2 open-label extension.

ELIGIBILITY:
Inclusion Criteria:

* Evidence of signed and dated informed consent document(s) indicating that the study candidate (and/or a parent/legal guardian) has been informed of all pertinent aspects of the study. Note: If the study candidate is considered a child under local regulation, a parent or legal guardian must provide written consent prior to initiation of study screening procedures and the study candidate may be required to provide written assent. The rules of the responsible institutional review board/independent ethics committee (IRB/IEC) regarding whether 1 or both parents must provide consent and the appropriate ages for obtaining consent and assent from the participant should be followed.
* Body weight greater than or equal to (>=) 12 kg.
* Documentation of the presence of a nonsense mutation in 1 allele of the PAX6 gene as determined by genotyping performed at a laboratory certified by the College of American Pathologists (CAP), or under the Clinical Laboratory Improvement Act/Amendment (CLIA), or by an equivalent organization.
* Clinical diagnosis of aniridia.
* Willingness and ability to comply with scheduled visits, drug administration plan, study procedures, and study restrictions.
* Good general health, as determined at Screening by medical history and physical examination (including vital sign measurements).
* No clinically significant abnormality based upon laboratory assessments at Screening, in the opinion of the investigator.
* Female participants of childbearing potential are eligible for the study but must be willing to use adequate (at least 1 form of) contraceptive methods as described below during the study treatment period (starting from the day of first dose of study drug and ending 60 days after the last dose of study drug). Childbearing potential is defined as participants who have experienced menarche and who are neither postmenopausal nor have been permanently sterilized.

  1. Hormonal methods of contraception (including oral and transdermal contraceptives, injectable progesterone, progestin subdermal implants, progesterone-releasing intrauterine devices [IUDs]) initiated at least 14 days prior to the first dose of study drug
  2. Abstinence
  3. Placement of a copper-containing IUD
  4. Condom with spermicidal foam/gel/film/cream/suppository
  5. Postmenopausal at least 12 months prior to first dose of study drug or permanently sterilized (for example, tubal occlusion, hysterectomy, bilateral salpingectomy)
  6. Male partner who has had a vasectomy for at least 3 months prior to the first dose of study drug
* Male participants with partners of childbearing potential must agree to use adequate (at least 1 form of) contraception as described below during the study treatment period (starting from the day of first dose of study drug and ending 60 days after the last dose of study drug).

  1. Abstinence
  2. Vasectomy for at least 3 months prior to first dose of study drug or surgically sterile
  3. Without a vasectomy, must use a condom with spermicidal foam/gel/film/cream suppository

Exclusion Criteria:

* Participants participating in any drug or device clinical investigation within 90 days prior to Screening or who anticipate participating in any other drug or device clinical investigation within the duration of this study.
* Exposure to ataluren within 90 days prior to Screening.
* Surgery within 30 days prior to enrollment.
* Female participants who are pregnant or breastfeeding. Female participants of childbearing potential must have a negative pregnancy test (beta-human chorionic gonadotropin [beta-HCG]) at screening and must use adequate (at least 1 form of) contraceptive methods.
* Active ocular infection or inflammation.
* Prior or ongoing medical condition (for example, concomitant illness, alcoholism, drug abuse, psychiatric condition), medical history, physical findings, or laboratory abnormality that, in the investigator's opinion, could adversely affect the safety of the participant, makes it unlikely that the course of study drug administration or follow-up would be completed, or could impair the assessment of study results.
* Participants with a positive result for hepatitis B, hepatitis C, or human immunodeficiency virus at Visit 1 (Screening).
* Ongoing warfarin, phenytoin, or tolbutamide therapy.
* Ongoing intravenous (IV) aminoglycoside or IV vancomycin use.
* Ongoing systemic cyclosporine therapy. Note: Topical cyclosporine therapy is permitted.
* Known hypersensitivity to any of the ingredients or excipients of the study drug (polydextrose, polyethylene glycol 3350, poloxamer 407, mannitol 25C, crospovidone XL10, hydroxyethyl cellulose, vanilla, colloidal silica, or magnesium stearate).
* 20/200 or worse visual acuity in the better eye with best correction.
* Participants who are monocular.
* Participants with a history of complications due to ocular surgery that could interfere with the study procedures or assessment of study endpoints.
* Participants with any other significant ocular or systemic disease that the Investigator determines could interfere with the study.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2016-01-31 (Actual); Primary Completion 2021-01-22 (Actual); Study Completion 2021-01-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Quintus Ngumah, OD, PhD, Study Director — PTC Therapeutics
Locations (3):
- United States (2):
  - Casey Eye Institute, Oregon Health & Science University, Portland, Oregon
  - University of Virginia, Charlottesville, Virginia
- University of British Columbia, Vancouver, British Columbia, Canada

RESULTS

PARTICIPANT FLOW:
Groups:
- Ataluren: Participants received ataluren orally 3 times a day (TID) at a dose of 10 milligrams (mg)/kilogram (kg) in the morning, 10 mg/kg at midday, and 20 mg/kg in the evening for 48 weeks in Stage 1 (double-masked period) and for additional 96 weeks in Stage 2 (open-label extension period). Participants, who completed Stage 2 and agreed to continue in open-label sub-study, continued to receive ataluren treatment at same dose as mentioned above, for 96 weeks.
- Placebo: Participants received placebo matched to ataluren TID orally in the morning, at midday, and in the evening for 48 weeks in Stage 1 (double-masked period) and ataluren orally TID at a dose of 10 mg/kg in the morning, 10 mg/kg at midday, and 20 mg/kg in the evening for additional 96 weeks in Stage 2 (open-label extension period). Participants, who completed Stage 2 and agreed to continue in open-label sub-study, continued to receive ataluren treatment at same dose as mentioned above, for 96 weeks.
Period: Stage 1: Double-Masked Period (48 Weeks)
Arm/Group | Ataluren | Placebo
Started | 26 | 13
Received at Least 1 Dose of Study Drug | 26 | 13
Completed | 22 | 12
Not Completed | 4 | 1
Not completed — Non-compliance with study drug | 0 | 1
Not completed — Other than specified | 4 | 0
Period: Stage 2: Open-Label Extension (96 Weeks)
Arm/Group | Ataluren | Placebo
Started | 22 | 11 (1 participant completed Stage 1 but did not enter open-label part)
Completed | 12 | 7
Not Completed | 10 | 4
Not completed — Adverse Event | 2 | 1
Not completed — Other than specified | 8 | 3
Period: Open-Label Sub-Study (96 Weeks)
Arm/Group | Ataluren | Placebo
Started | 10 (2 participants completed open-label 144-weeks but did not enter open-label sub-study) | 7
Completed | 2 | 3
Not Completed | 8 | 4
Not completed — Lost to Follow-up | 1 | 0
Not completed — Other than specified | 7 | 4

BASELINE CHARACTERISTICS:
Population: The safety population included all randomized participants who received at least 1 dose of study drug.
Groups:
- Ataluren: Participants received ataluren orally TID at a dose of 10 mg/kg in the morning, 10 mg/kg at midday, and 20 mg/kg in the evening for 48 weeks in Stage 1 (double-masked period) and for additional 96 weeks in Stage 2 (open-label extension period). Participants, who completed Stage 2 and agreed to continue in open-label sub-study, continued to receive ataluren treatment at same dose as mentioned above, for 96 weeks.
- Total: Total of all reporting groups
Arm/Group | Ataluren | Placebo | Total
Number analyzed (Participants) | 26 | 13 | 39
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.1 (10.12) | 19.2 (19.43) | 15.8 (13.88)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 8 | 18
  Male | 16 | 5 | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 26 | 12 | 38
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 3 | 2 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 22 | 11 | 33
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Maximum Reading Speed of Oculus Unitas (OU) (Both Eyes) at Week 48, as Measured Using the Minnesota Low Vision Reading Test (MNREAD) Acuity Charts
Description: MNREAD Acuity Chart can only be used to assess participants ≥8 years old. MNREAD Acuity Chart measures reading speed as a function of print size in participants with normal and low vision. The test consists of short sentences with print size decreasing by 0.1 log unit steps from a maximum of 1.3 logarithm of the minimum angle of resolution (logMAR) (equivalent to 20/400 or 6/120 when viewed at 40 centimeters [cm]) to -0.5 logMAR (equivalent to 20/6 or 6/2). An MNREAD Acuity Chart curve of reading speed vs print size has a typical shape for normally sighted persons and many low-vision individuals. This curve is characterized by 3 summary values. At large print sizes, reading speed remains fairly constant, forming a plateau that represents the maximum reading speed. As the print size decreases, a critical print size (CPS) is reached at which reading speed begins to decline rapidly. Finally, the smallest print size that can be read is defined as the reading acuity (RA).
Time Frame: Baseline, Week 48
Population: The intent-to-treat (ITT) population included all randomized participants who received at least 1 dose of study drug. Here, 'Overall number of participants analyzed' = participants evaluable for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Ataluren | Placebo
Number analyzed (Participants) | 11 | 5
percent change | 9.87 (7.425) | -0.89 (11.809)
Statistical Analysis 1: Comparison: Ataluren vs Placebo; Analysis was performed using analysis of covariance (ANCOVA) with age and baseline Maximum Reading Speed (both eyes) as covariates, and treatment as a factor; Test type: Other; p = 0.4868, ANCOVA — Threshold for significance at 0.05 level; Least Square (LS) Mean Difference = 10.76, 95% CI 2-sided [-21.914 to 43.434]

2. Secondary Outcome: Change From Baseline in Reading Accessibility Index of Both Eyes at Week 48
Description: Reading Accessibility Index is defined as the mean reading speed in words per minute (wpm) across the 10 largest physical print sizes on the MNREAD Acuity Chart, normalized by the value for a group of normally sighted young adults. For a viewing distance of 40 cm, this range of print sizes corresponds to 0.4 to 1.3 logMAR. This range of print sizes was chosen for 2 reasons. First, it sustains the manifest refraction spherical equivalent (MRS) in normally sighted persons. Second, it covers most contemporary printed text found in everyday life. Because the Reading Accessibility Index is normalized by the value for a group of normally sighted young adults (aged 18 to 39 years), a Reading Accessibility Index of 1.0 represents normal performance for this age group. Values less than 1.0 mean reduced accessibility to printed text within the range of print size encountered in daily life. Missing data was imputed using last observation carried forward (LOCF) method.
Time Frame: Baseline, Week 48
Population: The ITT population included all randomized participants who received at least 1 dose of study drug. Here, 'Overall number of participants analyzed' = participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ataluren | Placebo
Number analyzed (Participants) | 11 | 6
units on a scale | 0.10 (0.241) | 0.02 (0.267)

3. Secondary Outcome: Change From Baseline in Best Corrected Visual Acuity (BCVA) at Week 48
Description: The BCVA was evaluated using the Early Treatment Diabetic Retinopathy Study (ETDRS) Method. Missing data was imputed using LOCF method.
Time Frame: Baseline, Week 48
Population: The ITT population included all randomized participants who received at least 1 dose of study drug. Here, 'Overall number of participants analyzed' = participants evaluable for this outcome measure. 'Number analyzed' = participants evaluable for specified category.
Measure: Mean (Standard Deviation); unit: LogMAR
Arm/Group | Ataluren | Placebo
Number analyzed (Participants) | 24 | 13
LogMAR
  Left Eye: number analyzed (Participants) | 22 | 13
  Left Eye | -0.00 (0.076) | 0.01 (0.103)
  Right Eye | 0.03 (0.125) | -0.04 (0.138)

4. Secondary Outcome: Percent Change From Baseline in Maximum Reading Speed of Oculus Dexter (OD) (Right Eye) and Oculus Sinister (OS) (Left Eye) at Week 48
Description: Maximum Reading Speed was measured using the MNREAD Acuity Chart, which can only be used to assess participants ≥8 years old. The MNREAD Acuity Chart measures reading speed as a function of print size in participants with normal and low vision. The test consists of short sentences with print size decreasing by 0.1 log unit steps from a maximum of 1.3 logMAR (equivalent to 20/400 or 6/120 when viewed at 40 cm) to -0.5 logMAR (equivalent to 20/6 or 6/2). An MNREAD Acuity Chart curve of reading speed vs print size has a typical shape for normally sighted persons and many low-vision individuals. This curve is characterized by 3 summary values. At large print sizes, reading speed remains fairly constant, forming a plateau that represents the maximum reading speed. As the print size decreases, a CPS is reached at which reading speed begins to decline rapidly. Finally, the smallest print size that can be read is defined as the RA.
Time Frame: Baseline, Week 48
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Ataluren | Placebo
Number analyzed (Participants) | 10 | 6
percent change
  Left Eye: number analyzed (Participants) | 10 | 4
  Left Eye | 8.70 (36.464) | -4.11 (38.380)
  Right Eye: number analyzed (Participants) | 8 | 6
  Right Eye | 19.05 (39.116) | -3.83 (21.091)

5. Secondary Outcome: Change From Baseline in Reading Accessibility Index of Right Eye and Left Eye at Week 48
Description: Reading Accessibility Index is defined as the mean reading speed in wpm across the 10 largest physical print sizes on the MNREAD Acuity Chart, normalized by the value for a group of normally sighted young adults. For a viewing distance of 40 cm, this range of print sizes corresponds to 0.4 to 1.3 logMAR. This range of print sizes was chosen for 2 reasons. First, it sustains the MRS in normally sighted persons. Second, it covers most contemporary printed text found in everyday life. Because the Reading Accessibility Index is normalized by the value for a group of normally sighted young adults (aged 18 to 39 years), a Reading Accessibility Index of 1.0 represents normal performance for this age group. Values less than 1.0 mean reduced accessibility to printed text within the range of print size encountered in daily life. Missing data was imputed using LOCF method.
Time Frame: Baseline, Week 48
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ataluren | Placebo
Number analyzed (Participants) | 11 | 6
units on a scale
  Left Eye: number analyzed (Participants) | 11 | 4
  Left Eye | -0.70 (2.601) | 0.01 (0.224)
  Right Eye: number analyzed (Participants) | 9 | 6
  Right Eye | 0.04 (0.048) | 0.05 (0.128)

6. Secondary Outcome: Change From Baseline in Critical Print Size (CPS) of Both Eyes, Right Eye, and Left Eye at Week 48
Description: The MNREAD Acuity Chart measures reading speed as a function of print size in participants with normal and low vision. The test consists of short sentences with print size decreasing by 0.1 log unit steps from a maximum of 1.3 logMAR (equivalent to 20/400 or 6/120 when viewed at 40 cm) to -0.5 logMAR (equivalent to 20/6 or 6/2). An MNREAD Acuity Chart curve of reading speed vs print size has a typical shape for normally sighted persons and many low-vision individuals. This curve is characterized by 3 summary values. At large print sizes, reading speed remains fairly constant, forming a plateau that represents the maximum reading speed. As the print size decreases, a CPS is reached at which reading speed begins to decline rapidly. Finally, the smallest print size that can be read is defined as the RA. Missing data was imputed using LOCF method.
Time Frame: Baseline, Week 48
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: LogMAR
Arm/Group | Ataluren | Placebo
Number analyzed (Participants) | 11 | 6
LogMAR
  Both Eyes | -0.19 (0.259) | 0.12 (0.433)
  Left Eye: number analyzed (Participants) | 10 | 4
  Left Eye | -0.05 (0.198) | 0.07 (0.271)
  Right Eye: number analyzed (Participants) | 9 | 6
  Right Eye | 0.03 (0.275) | -0.02 (0.452)

7. Secondary Outcome: Change From Baseline in Reading Acuity (RA) of Both Eyes, Right Eye, and Left Eye at Week 48
Description: as for outcome 6
Time Frame: Baseline, Week 48
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: LogMAR
Arm/Group | Ataluren | Placebo
Number analyzed (Participants) | 11 | 6
LogMAR
  Both Eyes | -0.06 (0.239) | -0.16 (0.339)
  Left Eye: number analyzed (Participants) | 11 | 4
  Left Eye | -0.15 (2.723) | -0.16 (0.467)
  Right Eye: number analyzed (Participants) | 9 | 6
  Right Eye | -0.05 (0.142) | -0.14 (0.236)

8. Secondary Outcome: Number of Participants With Change From Baseline in Severity of Corneal Keratopathy at Week 48
Description: The severity of corneal keratopathy was reported as worsened, not change, or improve. Missing data were imputed using LOCF.
Time Frame: Baseline to Week 48
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Ataluren | Placebo
Number analyzed (Participants) | 21 | 12
Participants
  Left Eye: number analyzed (Participants) | 19 | 7
  Left Eye: Worsened | 4 | 2
  Left Eye: Not change | 7 | 2
  Left Eye: Improved | 8 | 3
  Right Eye: number analyzed (Participants) | 21 | 8
  Right Eye: Worsened | 4 | 2
  Right Eye: Not change | 7 | 2
  Right Eye: Improved | 10 | 4

9. Secondary Outcome: Change From Baseline in Iris Area at Week 48
Description: Missing data were imputed using LOCF.
Time Frame: Baseline, Week 48
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: millimeter square (mm^2)
Arm/Group | Ataluren | Placebo
Number analyzed (Participants) | 9 | 2
millimeter square (mm^2)
  Left Eye: number analyzed (Participants) | 6 | 2
  Left Eye | -0.15 (0.333) | 0.14 (0.129)
  Right Eye: number analyzed (Participants) | 9 | 1
  Right Eye | -0.06 (0.257) | -0.14

10. Secondary Outcome: Change From Baseline in BCVA at Week 240
Description: The BCVA was evaluated using the ETDRS Method. Missing data were imputed using LOCF method.
Time Frame: Baseline, Week 240
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | Ataluren | Placebo
Number analyzed (Participants) | 2 | 0
logMAR
  Left Eye | 0.02 (0.141) |
  Right Eye | 0.11 (0.240) |

11. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. AEs included both SAEs and non-serious AEs. A summary of other non-serious AEs and all SAEs, regardless of causality is located in the 'Reported AE section'. AEs were summarized separately for Stage 1 and for the overall ataluren experience, which included all participants who received ataluren throughput the study (Stage 1, open-label extension period [Stage 2], and sub-study).
Time Frame: Baseline up to Week 244
Population: The safety population included all randomized participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Groups:
- Stage 1: Ataluren: Participants received ataluren orally TID at a dose of 10 mg/kg in the morning, 10 mg/kg at midday, and 20 mg/kg in the evening for 48 weeks in Stage 1 (double-masked period).
- Stage 1: Placebo: Participants received placebo matched to ataluren TID orally in the morning, at midday, and in the evening for 48 weeks in Stage 1 (double-masked period).
- Overall Ataluren Exposure: Participants received ataluren orally TID at a dose of 10 mg/kg in the morning, 10 mg/kg at midday, and 20 mg/kg in the evening for 48 weeks in Stage 1 (double-masked period) and for additional 96 weeks in Stage 2 (open-label extension period). Participants, who completed Stage 2 and agreed to continue in open-label sub-study, continued to receive ataluren treatment at same dose as mentioned above, for 96 weeks.
Arm/Group | Stage 1: Ataluren | Stage 1: Placebo | Overall Ataluren Exposure
Number analyzed (Participants) | 26 | 13 | 37
Participants | 22 | 10 | 35

ADVERSE EVENTS:
Time Frame: Baseline up to Week 244
Description: The safety population included all randomized participants who received at least 1 dose of study drug. AEs were summarized separately for Stage 1 and for the overall ataluren experience, which included all participants who received ataluren throughput the study (Stage 1, open-label extension period [Stage 2], and sub-study).
Arm/Group | Stage 1: Ataluren | Stage 1: Placebo | Overall Ataluren Exposure
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/13 | 0/37
Serious Adverse Events (participants affected / at risk) | 1/26 | 0/13 | 1/37
Other Adverse Events (participants affected / at risk) | 22/26 | 10/13 | 35/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Stage 1: Ataluren (N=26) | Stage 1: Placebo (N=13) | Overall Ataluren Exposure (N=37)
Mental disorder (Psychiatric disorders) | 1 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Stage 1: Ataluren (N=26) | Stage 1: Placebo (N=13) | Overall Ataluren Exposure (N=37)
Abdominal pain upper (Gastrointestinal disorders) | 5 | 3 | 9
Vomiting (Gastrointestinal disorders) | 5 | 3 | 8
Nausea (Gastrointestinal disorders) | 4 | 2 | 4
Flatulence (Gastrointestinal disorders) | 3 | 1 | 3
Abdominal distension (Gastrointestinal disorders) | 2 | 1 | 2
Frequent bowel movements (Gastrointestinal disorders) | 2 | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 2
Dental caries (Gastrointestinal disorders) | 1 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 2
Faeces soft (Gastrointestinal disorders) | 1 | 0 | 1
Tooth impacted (Gastrointestinal disorders) | 1 | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 0 | 2 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 1
Gastrointestinal Pain (Gastrointestinal disorders) | 0 | 0 | 1
Malaise (General disorders) | 5 | 2 | 9
Fatigue (General disorders) | 1 | 0 | 1
Local swelling (General disorders) | 1 | 0 | 1
Medical device site reaction (General disorders) | 1 | 0 | 1
Pyrexia (General disorders) | 1 | 1 | 6
Asthenia (General disorders) | 0 | 1 | 0
Sensation of pressure (General disorders) | 0 | 1 | 0
Pain (General disorders) | 0 | 0 | 1
Dry eye (Eye disorders) | 4 | 3 | 9
Lacrimation increased (Eye disorders) | 3 | 1 | 10
Eye pruritus (Eye disorders) | 2 | 2 | 13
Corneal opacity (Eye disorders) | 1 | 0 | 1
Eye swelling (Eye disorders) | 1 | 0 | 1
Eyelid ptosis (Eye disorders) | 1 | 0 | 1
Lenticular opacities (Eye disorders) | 1 | 0 | 1
Ocular hyperaemia (Eye disorders) | 1 | 0 | 2
Eye discharge (Eye disorders) | 0 | 2 | 3
Keratopathy (Eye disorders) | 0 | 1 | 1
Vision blurred (Eye disorders) | 0 | 1 | 1
Vitreous detachment (Eye disorders) | 0 | 1 | 0
Photophobia (Eye disorders) | 0 | 0 | 17
Eye pain (Eye disorders) | 0 | 0 | 4
Lens discolouration (Eye disorders) | 0 | 0 | 2
Blepharospasm (Eye disorders) | 0 | 0 | 1
Cataract (Eye disorders) | 0 | 0 | 1
Eye inflammation (Eye disorders) | 0 | 0 | 1
Eye irritation (Eye disorders) | 0 | 0 | 1
Photokeratitis (Eye disorders) | 0 | 0 | 1
Punctate keratitis (Eye disorders) | 0 | 0 | 1
Visual acuity reduced (Eye disorders) | 0 | 0 | 1
Gastroenteritis viral (Infections and infestations) | 2 | 0 | 7
Conjunctivitis (Infections and infestations) | 1 | 0 | 5
Influenza (Infections and infestations) | 1 | 0 | 6
Nasopharyngitis (Infections and infestations) | 1 | 1 | 1
Pharyngitis streptococcal (Infections and infestations) | 1 | 0 | 2
Roseola (Infections and infestations) | 1 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 1
Ear infection (Infections and infestations) | 0 | 1 | 0
Atypical Pneumonia (Infections and infestations) | 0 | 0 | 1
Cellulitis of male external genital organ (Infections and infestations) | 0 | 0 | 1
Eye infection (Infections and infestations) | 0 | 0 | 1
Lyme disease (Infections and infestations) | 0 | 0 | 1
Respiratory tract infection (Infections and infestations) | 0 | 0 | 1
Urine leukocyte esterase positive (Investigations) | 2 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0 | 2
Upper respiratory tract infection (Investigations) | 1 | 0 | 0
Blood uric acid increased (Investigations) | 1 | 0 | 2
Nitrite urine present (Investigations) | 1 | 0 | 1
Protein urine present (Investigations) | 1 | 0 | 1
Urine ketone body present (Investigations) | 1 | 0 | 1
Blood urea increased (Investigations) | 0 | 0 | 2
Intraocular pressure increased (Investigations) | 0 | 0 | 2
Urine Leukocyte esterase positive (Investigations) | 0 | 0 | 2
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 1
Bacterial test positive (Investigations) | 0 | 0 | 1
Blood bilirubin increased (Investigations) | 0 | 0 | 1
Hepatic enzyme increased (Investigations) | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 1 | 0 | 1
Mood altered (Psychiatric disorders) | 1 | 0 | 1
Attention deficit/Hyperactivity disorder (Psychiatric disorders) | 0 | 0 | 2
Anxiety (Psychiatric disorders) | 0 | 0 | 1
Depression (Psychiatric disorders) | 0 | 0 | 1
Obsessive-compulsive disorder (Psychiatric disorders) | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 2 | 0 | 2
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Hypothyroidism (Endocrine disorders) | 1 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 1
Somnolence (Nervous system disorders) | 1 | 0 | 1
Headache (Nervous system disorders) | 0 | 1 | 3
Migraine (Nervous system disorders) | 0 | 0 | 3
Concussion (Injury, poisoning and procedural complications) | 0 | 0 | 1
Corneal Abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 0 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 1
Radius fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Sunburn (Injury, poisoning and procedural complications) | 0 | 0 | 1
Haematuria (Renal and urinary disorders) | 1 | 0 | 1
Dysuria (Renal and urinary disorders) | 0 | 0 | 1
Epiphysiolysis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Menorrhagia (Reproductive system and breast disorders) | 0 | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Balanoposthitis (Reproductive system and breast disorders) | 0 | 0 | 1
Metrorrhagia (Reproductive system and breast disorders) | 0 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Phimosis (Congenital, familial and genetic disorders) | 0 | 0 | 1
Motion sickness (Ear and labyrinth disorders) | 0 | 0 | 1
Seasonal allergy (Immune system disorders) | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor can review results and/or communications prior to public release and can embargo communications regarding trial results for a period that is up to 180 days from the time submitted to the sponsor for review. The sponsor may consult with the PI to require changes to the communication or extend the embargo.

DOCUMENTS (2):
  • Study Protocol (2019-12-17): https://cdn.clinicaltrials.gov/large-docs/59/NCT02647359/Prot_000.pdf
  • Statistical Analysis Plan (2020-02-05): https://cdn.clinicaltrials.gov/large-docs/59/NCT02647359/SAP_001.pdf